CLINICAL TRIAL: NCT05942612
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-2001 After a Single or Multiple Subcutaneous Injections in Healthy Subjects
Brief Title: A Phase I Study of SHR -2001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-2001-101
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Cohort 1 (Experimental): A single subcutaneous injection of SHR-2001/placebo dose 1 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 2 (Experimental): A single subcutaneous injection of SHR-2001/placebo dose 2 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 3 (Experimental): A single subcutaneous injection of SHR-2001/placebo dose 3 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 4 (Experimental): A single subcutaneous injection of SHR-2001/placebo dose 4 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 5 (Experimental): A single subcutaneous injection of SHR-2001/placebo dose 5 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 6 (Experimental): A single subcutaneous injection of SHR-2001/placebo dose 6 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 7 (Experimental): A single subcutaneous injection of SHR-2001/placebo dose 7 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 8 (Experimental): A single subcutaneous injection of SHR-2001 / placebo dose 8 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 9 (Experimental): A single subcutaneous injection of SHR-2001 / placebo dose 9 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 10 (Experimental): A single subcutaneous injection of SHR-2001 / placebo dose 10 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 11 (Experimental): A multiple subcutaneous injection of SHR-2001 / placebo dose 11 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo
- Cohort 12 (Experimental): A multiple subcutaneous injection of SHR-2001 / placebo dose 12 in healthy subjects.
  Interventions: Drug: SHR-2001; Drug: Placebo

INTERVENTIONS:
Drug: SHR-2001 — Subcutaneous injection, single dose or multiple doses.
Drug: Placebo — Subcutaneous injection, single dose or multiple doses.

SUMMARY:
This study is a phase 1 single dose or multiple doses escalation study of SHR-2001 in healthy subjects. The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR-2001 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain informed consent from participants before the start of any study related activities. Participants must have a full understanding of the purpose and significance of the trial, and be willing to comply with the trial protocol;
2. Age 18 ~ 55 years old (including boundary value), male or female;
3. Weight ≥ 45 kg, body mass index (BMI) ranging 19 ~ 28 kg/m2 (including boundary value);
4. Participants who are overtly healthy as determined by medical history and physical examination.;
5. Participants and their partners have no fertility plan and voluntarily use highly effective contraception. Female subjects must have a negative serum pregnancy test and be non-lactating.

Exclusion Criteria:

1. Those who have serious systemic diseases within 3 months before screening or administration, and the investigator believes that there may be safety risks;
2. Those who have serious infection, severe trauma or major surgery within 6 months before screening or administration; those who plan to undergo surgery during the trial;
3. Inactivated vaccine received within 2 weeks prior to randomization or live attenuated vaccine within 3 months prior to randomization, or intended to be vaccinated during the study period;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 64 days).
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-t | Start of Treatment to end of study (approximately 64 days).
  Area under the concentration-time curve from 0 to the last measurable time point after SHR-2001 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 64 days).
  Area under the concentration-time curve from time 0 to infinity after SHR-2001 administration
Pharmacokinetics-Cmax | Start of Treatment to end of study (approximately 64 days).
  Maximum observed concentration of SHR-2001
Pharmacokinetics-Tmax | Start of Treatment to end of study (approximately 64 days).
  Time to Cmax
Pharmacokinetics-t1/2 | Start of Treatment to end of study (approximately 64 days).
  Terminal elimination half-life of SHR-2001
Pharmacokinetics-CL/F | Start of Treatment to end of study (approximately 64 days).
  Apparent clearance of SHR-2001
Pharmacokinetics-Vz/F | Start of Treatment to end of study (approximately 64 days).
  Apparent volume of distribution during terminal phase of SHR-2001
Anti-Drug antibody | Start of Treatment to end of study (approximately 64 days).
  The percentage of subjects with positive ADA

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided